CLINICAL TRIAL: NCT03938116
Title: Healing Hearts Together: Evaluating a Couples-based Intervention to Improve Health Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190101-01H
Record Dates: First submitted 2019-04-25; First posted 2019-05-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases
Keywords: couple relationship; heart disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healing Hearts Together (Experimental)
  Interventions: Other: Healing Hearts Together
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Healing Hearts Together — Participants in the HHT group will be assembled in groups and attend 8 weekly 2-hr sessions at UOHI led by 2 facilitators with psychology training. Sessions: 1) focus on understanding love, attachment, and their relationship to heart health; 2) provide an opportunity to share experiences related to cardiovascular disease with partners and peers; and 3) assist in identifying and improving communication patterns that may inhibit positive interactions and healthy behaviours. Participants are introduced to concepts through didactic presentations, videos, group and couple discussion and homework exercises. Participants will receive a folder containing copies of in-session and take-home exercises as well as the Hold Me Tight book to review between sessions.
  Arms: Healing Hearts Together

SUMMARY:
The purpose of this study is to test the efficacy of the 8-week Healing Hearts Together (HHT) program to improve relationship quality, mental health, quality of life (QoL), and cardiovascular health. This is a randomized controlled trial in which couples are randomly assigned to the HHT group or usual care. Changes in the outcomes of interest will be assessed at the end of the intervention (8 weeks) and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

1. University of Ottawa Heart Institute (UOHI) patients and their partners
2. Participants in a romantic relationship who are cohabiting (married, common-law or committed relationship for ≥1 year). No restrictions will be placed on sexual orientation.
3. Participants are ≥ 18 years of age
4. Participants are able to read and understand English (HHT materials are only available in English; once efficacy has been established, all materials will be translated to French).
5. Patients and partners are available to participate for the next 6 months (intervention and follow-up).
6. Patients and partners are able to provide informed consent.

Exclusion Criteria:

1. Participants who, in the opinion of the study psychologist, manifest psychiatric illness or cognitive impairment that would preclude participation in HHT (i.e. unable to benefit from the intervention; to prevent disruption of other participants).
2. Participants who are engaging in couples therapy or plan to engage in couples therapy in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Relationship quality: DAS | 8 weeks
  Relationship quality will be assessed using the DAS. The DAS is a validated 32-item questionnaire that measures couple satisfaction, cohesion, consensus and affectionate expression. Scores ≥108 are indicative of couple satisfaction, while scores ≤107 indicate distress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada